CLINICAL TRIAL: NCT06946823
Title: Community-Engaged Design and Implementation of a Just-In-Time Adaptive Intervention (JITAI) to Improve Adolescent Anxiety in Rural Populations
Brief Title: Implementation of a Just-In-Time Adaptive Intervention for Adolescent Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Elizabeth L. Murnane, Assistant Professor of Engineering, Trustees of Dartmouth College
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00033184
Record Dates: First submitted 2025-04-08; First posted 2025-04-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Anxiety Disorders; Anxiety Disorder of Childhood
Keywords: Anxiety; Just-In-Time Adaptive Intervention; Smartphone; Behavioral Health; Community-Engaged Research; Adolescents; Rural; Digital Intervention; Participatory Design; Somatic
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 50 rural adolescents experiencing elevated anxiety levels will be randomly assigned to the JITAI tool for a treatment period of 3 months or a waitlist control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Just-In-Time Adaptive Intervention for Adolescent Anxiety (Experimental): Participants in the Just-In-Time Adaptive Intervention for Adolescent Anxiety Arm will receive the just-in-time adaptive smartphone tool and be instructed to respond to the tool's prompts and follow delivered behavioral recommendations throughout the 3-month intervention period.
  Interventions: Device: Just-In-Time Adaptive Intervention for Adolescent Anxiety
- Waitlist Control (No Intervention): Participants in the Waitlist Control Arm will receive the just-in-time adaptive smartphone tool following the completion of the 3-month intervention period.

INTERVENTIONS:
Device: Just-In-Time Adaptive Intervention for Adolescent Anxiety — A JITAI smartphone app to reduce anxiety levels among rural adolescents by delivering somatic-based activity recommendations
  Arms: Just-In-Time Adaptive Intervention for Adolescent Anxiety

SUMMARY:
The goal of this clinical trial is to evaluate a smartphone based just-in-time adaptive intervention (JITAI) tool to deliver somatic behavioral recommendations for anxiety management among youth. The main questions it aims to answer are:

* Is the JITAI tool acceptable among the adolescent study population?
* Is the JITAI tool feasible to deliver to the adolescent study population?
* Does the study support preliminary efficacy of the JITAI tool among the adolescent study population?

The tool will be pilot-tested among a sample of 50 rural adolescents experiencing elevated anxiety levels who will be randomly assigned to the JITAI tool or a waitlist control, for a treatment period of 3 months.

Participants will be asked to:

* Use the smartphone based JITAI tool which will deliver somatic behavioral recommendations intended to manage anxiety levels for a treatment period of 3 months
* Respond to the tool's prompts on a daily basis and follow the delivered behavioral recommendations
* Complete anxiety and interoception assessments at study start, study end (3 months), and one-month follow-up
* Complete usability and user experience instruments at study end (3 months)

DETAILED DESCRIPTION:
It is imperative to improve the inclusive reach of effective anxiety treatments for adolescents. Anxiety disorders are among the most common psychiatric conditions in adolescents yet they are largely undertreated, particularly in rural areas. Behavioral interventions are efficacious in reducing anxiety symptoms while providing individuals with a toolkit of knowledge, skills, and techniques that empower self-care. As anxiety disorders involve an interconnected relationship between psychological and physiological processes, behavioral interventions that combine mind-body practices are coming to be seen as a particularly powerful therapeutic approach. Such treatments can include physical exercises, expressive movements, and other activities that emphasize interoception, autonomic reactivity, and the role of the body in processing and regulating emotions. However, research is needed to tailor these somatic approaches to an adolescent population, more rigorously evaluate their efficacy in diverse settings, and enhance their accessibility in traditionally underserved communities. Further, it is key to ensure such interventions are responsive and available in real-time, considering in-the-moment support is a critical aspect of quality anxiety care. Mobile technology is a promising platform for delivering personalized behavioral interventions at-scale and on-demand, including through emerging designs like just-in-time adaptive intervention(JITAI). This project aims to design, develop, and test a smartphone based JITAI tool to deliver somatic behavioral recommendations to manage anxiety levels. It will use a community-engaged research approach that partners with adolescents. Following qualitative needfinding to understand anxiety experiences and care needs as well as participatory design of the digital intervention, the tool will be pilot tested with a sample of 50 rural adolescents experiencing elevated anxiety levels who will be randomly assigned to the JITAI tool or a waitlist control, for a treatment period of 3 months. Objectives include demonstrating the acceptability, feasibility, and preliminary efficacy of this intervention approach.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent (age 13-17 years old)
* New Hampshire resident
* Fluency in English
* Able to provide assent
* At least mild (≥5) anxiety based on the GAD-7 assessment

Exclusion Criteria:

* Under 13 years old
* Over 17 years old
* Not a New Hampshire resident
* Unable to provide assent
* Less than mild (<5) anxiety based on the GAD-7 assessment

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Symptoms of Generalized Anxiety at 3 Months | Baseline and 3 months
  Units on a scale measured through the GAD-7 (Generalized Anxiety Disorder-7) self-report questionnaire. Minimum score = 0, maximum score = 21, with a higher score indicating worse anxiety symptoms.
Change from Post-Treatment Symptoms of Generalized Anxiety to 1-month follow-up | Post-Treatment (3 months after baseline) and 1-month follow-up (4 months after baseline)
  Units on a scale measured through the GAD-7 (Generalized Anxiety Disorder-7) self-report questionnaire. Minimum score = 0, maximum score = 21, with a higher score indicating worse anxiety symptoms.
Change from Baseline in Interoceptive Awareness at 3 Months | Baseline and 3 months
  Units on a scale measured through the MAIA-Y (Multidimensional Assessment of Interoceptive Awareness for Youth) self-report questionnaire. Minimum score = 1, maximum score = 5, with higher scores indicating greater interoceptive awareness.
Change from Post-Treatment Interoceptive Awareness to 1-month follow-up | Post-Treatment (3 months after baseline) and 1-month follow-up (4 months after baseline)
  Units on a scale measured through the MAIA-Y (Multidimensional Assessment of Interoceptive Awareness for Youth) self-report questionnaire. Minimum score = 1, maximum score = 5, with higher scores indicating greater interoceptive awareness.

SECONDARY OUTCOMES:
Pragmatic and Hedonic User Experience | 3 months after baseline
  The AttrakDiff instrument assesses 4 dimensions of user experience (usability, stimulation, identity, and attractiveness) using a 7-point semantic differential scale where respondents choose between bipolar adjective pairs to produce an overall mean score. Minimum score = -3, maximum score = +3, where higher scores indicate a more usable and appealing tool.
Technology Engagement | 3 months after baseline
  The GiggleGauge instrument assesses user engagement through a self-report questionnaire with a binary ordinal scale. Minimum score = 5, maximum score = 10, where higher scores indicate a more engaging tool.
User Engagement | 3 months after baseline
  The User Engagement Scale (UES) instrument assesses user engagement with digital interventions through a self-report questionnaire on a 5-point Likert scale. Minimum score = 1, maximum score = 5, where higher scores indicate a more engaging tool.
Percentage of app-based intervention activities completed by participants | Baseline through 3-month treatment period
  Compliance will be assessed by calculating the percentage of assigned app-based intervention activities completed by each participant over the 3-month treatment period. Completion data will be automatically recorded by the app.
Number of participants who complete the study | End of treatment period (3 months after baseline)
  Retention will be defined as the number of participants who remain enrolled and complete all study procedures through the end of the treatment period at 3 months.

IPD SHARING:
Plan to Share IPD: No